CLINICAL TRIAL: NCT06220448
Title: Exploring the Epidemiology and Burden of Blunt Adrenal Gland Injury in the Context of Major Trauma
Brief Title: Blunt ADrenal Gland injUrY (BAD GUY) Project
Acronym: BADGUY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BD-2024
Record Dates: First submitted 2024-01-11; First posted 2024-01-24 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Trauma; Adrenal Gland Injury
Keywords: Trauma; blunt adrenal gland trauma; major trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BAGI: patients suffering from thoraco-abdominal blunt trauma with and without blunt adrenal gland injury

SUMMARY:
Type: retrospective observational multicenter trial. Population of interest: adult patients suffering from thoraco-abdominal trauma undergoing both non-operative and operative management.

Hypothesis: Adrenal gland injury is a rare finding after blunt thoracoabdominal trauma. Short-term outcomes of blunt adrenal gland injury (BAGI) described in literature are contradictory. Reports on the outcomes related to this injury are variable and consider heterogeneous populations of trauma patients Aim: This study aims to explore the burden related to BAGI in an homogeneous population of patients sustaining blunt thoraco-abdominal trauma treated in different institution

DETAILED DESCRIPTION:
Adrenal gland injury is a rare finding after blunt thoracoabdominal trauma. The diagnosis can be accurately made with CT scan in stable patients, whilst in unstable patients, the detection can often be made during surgery, in the post-operative setting or postmortem. Short-term outcomes of blunt adrenal gland injury (BAGI) described in literature are contradictory. Studies reported BAGI as a high mortality risk injury. On the other hand, according to further reports, the presence of a BAGI is not considered a marker of severe injury or associated with an increased mortality rate.

Evidences the from a large multicenter cohort of selected trauma patients are lacking.

The study hypothesis is that BAGI is related to patients with higher trauma severity and worse overall outcome. By exploring the clinical burden related to BAGI the investigators aim to determine if this is related to the anatomical location of the injured organ or if in addition an underlying undisclosed pato-physiological mechanism is present. The investigatorspropose an international multicenter analysis on the epidemiology and the burden of BAGI in the context of major trauma, exploring differences between BAGI and non-BAGI patients.

Primary endpoint:

• Relationship between trauma severity (Injury Severity Score) of thoraco-abdominal trauma patients with BAGI versus torso trauma patients without BAGI

Secondary endpoint:

• Organ Injury Scale of the blunt adrenal trauma(OIS), overall survival, ICU length of stay, overall length of stay

Methods:

Patients will be enrolled according to the reported criteria. The following variables will be considered: - Demographic (age, sex, comorbidities) - Mechanism of trauma - Trauma bay and surgical management - Trauma severity (ISS, NISS, OIS, AIS) - Need for ventilation (Y/N, timing) - Data on vasoactive support - Post trauma clinical and laboratory parameters - Mortality - Length of stay (ICU, hospital) All information of patients will be extracted from our dedicated Trauma Registry and personal informations will be removed according to data anonymization, and collected in an electronic database.

Data will be reported in accordance with Strengthening the Reporting of Observational studies in Epidemiology guidelines (STROBE) for observational studies.

Statistical analysis A 1:1 propensity score matching analysis will be performed based on sex, setting of the trauma, trauma mechanism, age, ASA classification, intentionality of the trauma, Glasgow coma scale and Revised Trauma Score. Following the propensity score matching patients included with and without BAGI will be compared using χ2 test for categorical variables and t-student test or Mann-Whitney test according to sample distribution for continuous variables

ELIGIBILITY:
Inclusion criteria:

* Age > 16 years old
* All patients with blunt thoraco-abdominal trauma

Exclusion criteria:

* TBI with AIS > 3
* Isolated TBI and Spinal cord injury
* Patients died in emergency department

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients presenting to ED diagnosed with acute appendicitis and eligible for laparoscopic appendectomy
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Injury Severity Score (ISS) | 120 days after trauma
  The Injury Severity Score (ISS) is an established medical score to assess trauma severity.It correlates with mortality, morbidity and hospitalization time after trauma. It is used to define the term major trauma. A major trauma (or polytrauma) is defined as the Injury Severity Score being greater than 15.The AIS Committee of the Association for the Advancement of Automotive Medicine (AAAM) designed and improves upon the scale.
  Injury Severity Score Minimum: 0 Maximum: 75 The risk of mortality and post trauma complications raises with increasing values in Injury Severity Score.

SECONDARY OUTCOMES:
Presence and number of thoraco-abdominal injuries | 120 days
  The presence of a specific organ injury per each thoraco-abdominal organ will be registered, defining the presence of an injury as a dichotomous variable (0 absent, 1 present)
Organ Injury Scale of the blunt adrenal trauma(OIS) | 120 days
  The presence of a blunt adrenal gland injury will be registered and classified following the America Association for Surgery of Trauma Organ Injury Scale classification as follow:
  I Contusion II Laceration involving only cortex (<2 cm) III Laceration extending into medulla (> 2 cm) IV >50% parenchymal destruction V Total parenchymal destruction (including massive intraparenchymal hemorrhage) Avulsion from blood supply
Overall survival | 120 days
  The final outcome of the patient at 120 days will be registered as a dichotomous variable (0 survived, 1 dead)
Overall length of stay | 120 days
  The length of stay in the hospital will be recorded considering it as the time frame, in days, from patient's admission to the emergency department to death or to the discharge to home or a rehabilitation service
Overall length of stay at ICU | 120 days
  The length of stay in the Intensive Care Unit will be recorded considering it as the time frame, in days, from patient's admission in the ICU to death or to the discharge to a surgical or medical ward

CONTACTS AND LOCATIONS:
Locations (1):
- ASST GOM Niguarda, Miano, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Undecided